CLINICAL TRIAL: NCT04795349
Title: New Techniques to evAlUate Response to neOadjuvant Treatments in bReast cAncer: Can Breast Surgery be Avoided
Brief Title: New Techniques to evAlUate Response to neOadjuvant Treatments in bReast cAncer (AURORA)
Acronym: AURORA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AURORA
Record Dates: First submitted 2021-02-25; First posted 2021-03-12 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-02

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Neoadjuvant chemotherapy; Magnetic Resonance Imaging; Contrast mammography; Elastography
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NAC Patients. (Experimental): Breast cancer patients after NAC completion, prior to surgery
  Interventions: Procedure: Vacuum-assisted breast biopsy

INTERVENTIONS:
Procedure: Vacuum-assisted breast biopsy — In those patients with a radiological complete response by all the radiological imaging methods, a stereotactic biopsy will be performed before surgery. After that, a comparison will be done between the results of the pre surgical biopsy and the definitive pathology of the specimen.

SUMMARY:
The role of neoadjuvant chemotherapy (NAC) in breast cancer is well established. Increasing rates of pathologic complete response (pCR) has increased de-escalation of surgical techniques. The objective of the study is to evaluate new radiologic techniques that can accurately detect complete response in order to eliminate breast surgery. . . Currently, there are several imaging techniques for NAC response assessment (magnetic resonance imaging -MRI-, mammography and ultrasound), with good correlation in partial response, but they lack power in predicting complete pathological response. The investigators propose to use IVIM (Intravoxel incoherent motion), Kurtosis (DKI by Diffusion Kurtosis imaging) and diffusion tensor image (DTI) in MRI, contrast enhancement mammography and shear wave elastography for the evaluation of the response to systemic treatment in breast cancer patients. In order to validate the technique, in those patients with a radiological complete response by all the radiological imaging methods, a vacuum-assisted biopsy will be performed before surgery. After that, a comparison will be done between the results of the pre surgical biopsy and the definitive pathology of the specimen. So the investigators can evaluate if patients with complete radiological response after NAC, can be spared breast surgery.

DETAILED DESCRIPTION:
The role of neoadjuvant chemotherapy (NAC) in breast cancer is well established. In inoperable patients at the time of diagnosis, the goal of NAC is to achieve a pathologic complete response (pCR) which has shown that it improves disease-free survival when compared to those cases with residual tumoral cells. Detection of the presence of residual disease is crucial for surgical planning; the ultimate goal would be to avoid surgery in those patients who achieve a pCR, though nowadays validated techniques with power enough to detect this residual disease are lacking.

Currently, several imaging techniques for NAC response assessment are being used (magnetic resonance imaging -MRI-, mammography and ultrasound), with good correlation in partial response, but they lack power in predicting complete pathological response; among them, nowadays the most accurate is MRI. In recent years, the use of the diffusion-enhanced images have been proposed for the quantitative characterization and for helping to improve the specificity of dynamic contrast study.

The investigators propose to use a bi-exponential model, IVIM (Intravoxel incoherent motion), which differentiates between microperfusion used by microvascular blood flow from the diffusion of water. Kurtosis (DKI by Diffusion Kurtosis imaging) which quantifies the deviation from the Gaussian pattern and diffusion tensor image (DTI) which provides information on the microstructure and pathophysiology tumor, presenting a statistically significant relationship with tumor cellularity. Preliminary studies have reported promising results for the evaluation of the early response to systemic treatment in breast cancer patients. Its utility for NAC response assessment in these patients will be analysed.

Recent studies have evaluated the application of contrast mammography in the assessment of the response to NAC, with MRI-like results. It is a faster and cheaper technique compared to MRI radiological evaluation of the response after NAC through this technique will be assessed and compared its results with the different techniques used in previous studies / in daily practice.

Shear wave elastography is a very useful tool for the quantitative assessment of the tissue hardness that is widely used for differentiating benign lesions from malignant ones. Nowadays some studies are investigating its usefulness in the assessment of the radiological evaluation after NAC, with promising results in terms of early evaluation. In this study, the elastography will be performed on pre surgical evaluation and its correlation with pathological anatomy.

In order to validate the technique, in those patients with a radiological complete response by all the radiological imaging methods, a stereotactic biopsy will be performed before surgery. After that, a comparison will be done between the results of the pre surgical biopsy and the definitive pathology of the specimen. If the false negative rate of the presurgical assessment including the biopsy are below 5%, patients could spare surgery when there is a complete radiological response. Objectives :

To evaluate if patients with complete radiological response after NAC, in this setting can be spared breast surgery. . - To determine if IVIM, KURTOSIS or DTI diffusion sequences in MRI can assess the response to NAC better than conventional sequences and, thus, be able to avoid the use of intravenous contrast in the MRI study in the future. - To determine whether the study of breast elastography with shear wave technology, is more sensitive or specific in the detection of residual tumor after NAC in breast cancer. - To determining whether contrast enhanced mammography helps us to assess the response to NAC in breast cancer, compared to MRI standard practice.

The expected results are:

False negative rate of pre-surgery biopsy <5%. Achieve a sensitivity >80% for the radiological tests in predicting pCR for selected tumoral subtypes (Triple Negative and HER2 enriched tumors).

Noninferiority of contrast mammography compared to breast MRI in determining the response to NAC.

ELIGIBILITY:
Inclusion Criteria:

* Women with Pathologic diagnosis of breast cancer with indication of neoadjuvant chemotherapy

Exclusion Criteria:

* Breast cancer recurrence
* Other synchronic tumour.
* Inflammatory cancer.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Complete Radiological Response | 6 months after NAC initiation
  To evaluate if patients with complete radiological response after NAC, in this setting can be spared breast surgery.

SECONDARY OUTCOMES:
MRI Measurements | 6 months after NAC initiation
  To determine if IVIM, KURTOSIS or DTI diffusion sequences in MRI can assess the response to NAC better than conventional sequences and, thus, be able to avoid the use of intravenous contrast in the MRI study in the future.
Elastography | 6 months after NAC initiation
  To determine whether the study of breast elastography with shear wave technology, is more sensitive or specific in the detection of residual tumor after NAC in breast cancer.
MRI Comparison | 6 months after NAC initiation
  To determining whether contrast enhanced mammography helps us to assess the response to NAC in breast cancer, compared to MRI standard practice.

CONTACTS AND LOCATIONS:
Locations (1):
- Clínica Universidad de Navarra, Madrid, Spain

REFERENCES:
- [Background] Heil J, Kuerer HM, Pfob A, Rauch G, Sinn HP, Golatta M, Liefers GJ, Vrancken Peeters MJ. Eliminating the breast cancer surgery paradigm after neoadjuvant systemic therapy: current evidence and future challenges. Ann Oncol. 2020 Jan;31(1):61-71. doi: 10.1016/j.annonc.2019.10.012. PMID 31912797
- [Background] Croshaw R, Shapiro-Wright H, Svensson E, Erb K, Julian T. Accuracy of clinical examination, digital mammogram, ultrasound, and MRI in determining postneoadjuvant pathologic tumor response in operable breast cancer patients. Ann Surg Oncol. 2011 Oct;18(11):3160-3. doi: 10.1245/s10434-011-1919-5. Epub 2011 Sep 27. PMID 21947594
- [Background] Marinovich ML, Houssami N, Macaskill P, Sardanelli F, Irwig L, Mamounas EP, von Minckwitz G, Brennan ME, Ciatto S. Meta-analysis of magnetic resonance imaging in detecting residual breast cancer after neoadjuvant therapy. J Natl Cancer Inst. 2013 Mar 6;105(5):321-33. doi: 10.1093/jnci/djs528. Epub 2013 Jan 7. PMID 23297042
- [Background] Sun K, Chen X, Chai W, Fei X, Fu C, Yan X, Zhan Y, Chen K, Shen K, Yan F. Breast Cancer: Diffusion Kurtosis MR Imaging-Diagnostic Accuracy and Correlation with Clinical-Pathologic Factors. Radiology. 2015 Oct;277(1):46-55. doi: 10.1148/radiol.15141625. Epub 2015 May 4. PMID 25938679
- [Background] Furman-Haran E, Nissan N, Ricart-Selma V, Martinez-Rubio C, Degani H, Camps-Herrero J. Quantitative evaluation of breast cancer response to neoadjuvant chemotherapy by diffusion tensor imaging: Initial results. J Magn Reson Imaging. 2018 Apr;47(4):1080-1090. doi: 10.1002/jmri.25855. Epub 2017 Sep 13. PMID 28901594
- [Background] Katyan A, Mittal MK, Mani C, Mandal AK. Strain wave elastography in response assessment to neo-adjuvant chemotherapy in patients with locally advanced breast cancer. Br J Radiol. 2019 Jul;92(1099):20180515. doi: 10.1259/bjr.20180515. Epub 2019 May 16. PMID 31045431